CLINICAL TRIAL: NCT05263752
Title: Evaluation of Safety and Efficacy of NvisionVLE® Imaging Low Profile System in Patients With Bile Duct Disease
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 059.GID.2017.D
Record Dates: First submitted 2019-08-12; First posted 2022-03-03 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Bile Duct Diseases
MeSH Terms: conditions — Bile Duct Diseases | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Undergone ERCP with NvisionVLE® Imaging Low Profile System: Undergone ERCP with NvisionVLE® Imaging Low Profile System at MDMC between 10/15/2017 and 10/15/2019
  Interventions: Device: ERCP with NvisionVLE® Imaging Low Profile System

INTERVENTIONS:
Device: ERCP with NvisionVLE® Imaging Low Profile System — Endoscopic Retrograde Cholangio-Pancreatography (ERCP) with NvisionVLE® Imaging Low Profile System

SUMMARY:
A previous study evaluating the NvisionVLE® Imaging Low Profile System revealed the system to be feasible and safe for use in bile duct. The study also revealed a potential to better define abnormalities, target sampling and therapy when utilizing the NvisionVLE® Imaging Low Profile System. This study will further evaluate the safety and efficacy of the NvisionVLE® Imaging Low Profile System in patients with bile duct diseases.

DETAILED DESCRIPTION:
The primary objective of this retrospective and prospective study is to acquire additional data to further evaluate the safety and efficacy of the NvisionVLE® Imaging Low Profile System in patients with bile duct disease. The secondary objective will be to provide a tool for participating physicians to collect imaging data, clinical utility data, and other clinical data such as demographics, pathology, and treatment surveillance results for patients who have undergone an examination of the bile duct with the NvisionVLE® Imaging Low Profile System. Specific aims include completing a multi-center registry to further evaluate the safety and efficacy of the NvisionVLE® Imaging System Low Profile System and developing a tool from the NvisionVLE® Imaging Low Profile System data to better define abnormalities, target sampling and therapy in patients with bile duct disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Undergone ERCP with NvisionVLE® Imaging Low Profile System at MDMC between 10/15/2017 and 10/15/2019.

Exclusion Criteria:

* Below 18 years of age
* Did not undergo ERCP with NvisionVLE® Imaging Low Profile System at MDMC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients over the age of 18 years who are scheduled to undergo an ERCP with Nvision VLE Imaging Low Profile System.
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Demographics- DOB | up to 2 years
  Date of birth
Demographics- Sex | up to 2 years
  Male/Female
Indication of Procedure | up to 2 years
  Anatomy Used: Biliary or Pancreatic
Previous Surgical History | up to 2 years
  Stent type and Location
Previous Imaging | up to 2 years
  Type of Imaging: CT or MRI for example
Previous Procedures | up to 2 years
  EUS or ERCP

CONTACTS AND LOCATIONS:
Overall Officials: Prashant Kedia, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Methodist Health System, Dallas, Texas, United States